CLINICAL TRIAL: NCT01864759
Title: Phase I Clinical Trial of Endovenous Administration of Conditionally Replicative Adenovirus ICOVIR-5 in Patients With Locally Advanced or Metastatic Melanoma
Brief Title: Phase I Endovenous Administration of Oncolytic Adenovirus ICOVIR-5 in Patients With Advanced or Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICOVIR5-2; 2008-005694-35 (EudraCT Number)
Record Dates: First submitted 2013-05-22; First posted 2013-05-30 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Locally Advanced or Metastatic Melanoma
Keywords: melanoma; oncolytic; adenovirus; virotherapy; locally advanced; metastatic
MeSH Terms: conditions — Melanoma; Adenoviridae Infections; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICOVIR5 (Experimental): ICOVIR-5 oncolytic adenovirus, single administration, endovenous, dose escalation from 1E11 vp to 1E13 vp.
  Interventions: Biological: ICOVIR-5

INTERVENTIONS:
Biological: ICOVIR-5

SUMMARY:
The investigators will evaluate the safety of a single endovenous infusion of ICOVIR5 in adults with locally advanced and metastatic melanoma. ICOVIR5 consists in a conditionally replicative or oncolytic adenovirus.

ELIGIBILITY:
Inclusion Criteria:

* Malignant melanoma advanced or metastatic.
* Other than 18 years
* Karnofsky index > 60 %
* Life expectancy > 3 months
* ALT/AST <=2.5 times the upper normal limit
* Creatinine clearance >= 50 ml/min.
* Bilirubin <25 umol/l
* Alkaline phosphatase <= 2.5 time upper normal limit
* Normal bone marrow function: Neutrophils >=1.5 E9/L, platelets >= 1E11/L, hemoglobin >= 100 g/l, Normal prothrombin time and thromboplastin time,
* HIV negative
* Measurable disease
* Signed informed consent.

Exclusion Criteria:

* Geographical, social or psychological conditions that may impair the protocol compliance.
* Active infections or other severe medical status.
* History of liver disease.
* Other or concomitant treatments for melanoma or investigational product.
* Previous participation in studies with adenovirus.
* Virus diseases diagnosed two weeks before inclusion.
* Immunosuppressive concomitant treatments
* Concomitant malignant haematological disease.
* Patients having family members with immunodeficient status or disease
* Patients with Li Fraumeni syndrome or germinal retinoblastoma gene defects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01-11 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 weeks
  The highest dose where less than two out of three or six patients suffered dose limiting toxicity.

SECONDARY OUTCOMES:
Recommended dose | 4 weeks
Anti-tumour activity | 4 weeks

OTHER OUTCOMES:
Viral pharmacokinetics | 1 day
  Viremia at 0 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours and 24 hours after endovenous injection.
Viral pharmacodynamics | 5 days
  Virus presence in tumors at day 5 post-administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Salazar, MD PhD, Principal Investigator — Institut Català d'Oncologia; Ramon Alemany, PhD, Study Chair — Institut Català d'Oncologia
Locations (1):
- Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet Del Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Cascallo M, Alonso MM, Rojas JJ, Perez-Gimenez A, Fueyo J, Alemany R. Systemic toxicity-efficacy profile of ICOVIR-5, a potent and selective oncolytic adenovirus based on the pRB pathway. Mol Ther. 2007 Sep;15(9):1607-15. doi: 10.1038/sj.mt.6300239. Epub 2007 Jun 19. PMID 17579575